CLINICAL TRIAL: NCT00985036
Title: Is VEGF a Useful Serum Biomarker for Patients Diagnosed With Meningioma or Glioma?
Brief Title: Vascular Endothelial Growth Factor (VEGF) Levels in Brain Tumor Patients
Status: Withdrawn | Type: Observational
Sponsor: Marquette General Health System (Other)
Collaborators: Upper Michigan Brain Tumor Center (Other)
Responsible Party: Principal Investigator, Richard A. Rovin, MD FACS, Neurosurgeon, Marquette General Health System
Other Study IDs: MGH-VEGF-1
Record Dates: First submitted 2009-09-25; First posted 2009-09-28 (Estimated); Last update posted 2012-04-24 (Estimated); Status verified 2012-04

CONDITIONS: Glioma; Meningioma
Keywords: glioma; meningioma; VEGF
MeSH Terms: conditions — Glioma; Meningioma | interventions — Hematologic Tests

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — serum
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Glioma: patients who are diagnosed with and are being treated for glioma
  Interventions: Procedure: Blood test
- meningioma: patients who are diagnosed with and are being treated for meningioma
  Interventions: Procedure: Blood test

INTERVENTIONS:
Procedure: Blood test — an additional vial of blood will be obtained at the time of MRI or at the time of routine blood tests ordered by the medical oncologist. In other words, there will be no extra needle sticks. Just an extra vial of blood will be taken during a routine blood test

SUMMARY:
Objectives: This study is looking at the level of vascular endothelial growth factor (VEGF) circulating in the blood stream of patients diagnosed with either a meningioma or a glioma. The questions that will be addressed include:

1. Can VEGF level alert us to tumor progression or recurrence before MRI changes occur?
2. Is the VEGF level an indicator of the response to treatment?
3. Does the VEGF level correlate with tumor histology and behavior?
4. Is there a relationship between VEGF level and outcome?

ELIGIBILITY:
Inclusion Criteria:

* any patient presenting with glioma or meningioma

Exclusion Criteria:

* a different type of brain tumor

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Patients presenting to Marquette General Hospital with a probable or confirmed diagnosis of meningioma or glioma
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2009-09; Primary Completion 2011-09 (Estimated); Study Completion 2012-01 (Estimated)

PRIMARY OUTCOMES:
Determine if VEGF levels correlate with tumor progression or recurrence | every one to three months

SECONDARY OUTCOMES:
Determine if the VEGF level is an indicator of the response to treatment. | Every one to three months
Determine if the VEGF level correlates with tumor histology and behavior. | Every one to three months
Determine if there is a relationship between VEGF level and outcome. | Every one to three months

CONTACTS AND LOCATIONS:
Overall Officials: Richard A Rovin, MD, FACS, Principal Investigator — Upper Michigan Brain Tumor Center; Robert J Winn, PhD, Principal Investigator — Northern Michigan University; Suresh Nukala, MD, Principal Investigator — Marquette General Health Systems
Locations (1):
- Marquette General Hospital, Marquette, Michigan, United States